CLINICAL TRIAL: NCT04857541
Title: Investigation of Breathing Performance of Healthy Young Adult
Brief Title: Breathing Performance of Healthy Young Adult
Status: Completed | Type: Observational
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Principal Investigator, Ching-Hsia Hung, Professor, National Cheng Kung University
Other Study IDs: A-ER-110-051
Record Dates: First submitted 2021-04-15; First posted 2021-04-23 (Actual); Last update posted 2022-06-10 (Actual); Status verified 2022-06

CONDITIONS: COPD; COPD-like
Keywords: COPD; Diaphragm; Voluntary cough; Abdominal muscle activation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Health adult

SUMMARY:
The study will recruit subject of healthy adult, COPD-like patient and patient with COPD to investigate the difference of respiratory performance. We will measure the body composition, respiratory muscle force, pulmonary function and performance of voluntary cough. The muscle thickness of abdominal muscle and diaphragm, assessment of diaphragm during different breathing pattern and the muscle activation during voluntary cough will also being determined. We hypothesized that there will be a significantly different between three group on the performance of voluntary cough, and the correlation between each variable will be further investigated.

DETAILED DESCRIPTION:
The specific aims of the study are:

1. difference of respiratory muscle performance between three groups
2. the correlation between respiratory symptom and pulmonary functional test
3. difference of functional respiratory performance (peak cough flow of voluntary cough) between three groups
4. muscle activation of abdominal muscle and diaphragm during performing voluntary force
5. performance of diaphragm under different breathing load

ELIGIBILITY:
1. Health subject

   Inclusion Criteria:
   * aged 20 years or above
   * currently not being diagnosis as COPD
   * less than 4 times/week of aerobic exercise
2. COPD-like subject

   Inclusion Criteria:
   * aged 20 years or above
   * currently not being diagnosis as COPD
   * presented of COPD symptoms (coughing, sputum production and dyspnea), last for 3 months and more than 2 years
   * score more than 1 on modified Medical Research Council (mMRC) or COPD Assessment Test (CAT)
3. COPD subject

Inclusion Criteria:

* aged 20 years or above
* currently being diagnosis as COPD
* haven't participated in any pulmonary rehabilitation program in the past three months

Exclusion Criteria:

* Untreated comorbidities for COPD
* Postural asymmetries (Scoliosis, length discrepancy of the lower limbs or other previous surgical history of spine)
* Chronic nonspecific lumbopelvic pain
* Gynecological or abdominal surgery in the previous year
* Pregnancy or post-delivery in the previous 6 months
* Neurological or inflammatory disorders
* Any conditions that may interfere with the data collection

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. Health subject: healthy adults with no existed respiratory condition
  2. COPD-like subject: subjects with COPD-like symptoms but not reach the diagnosis criteria
  3. COPD subject: subjects with diagnosed COPD
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2021-05-11 (Actual); Primary Completion 2021-05-13 (Actual); Study Completion 2022-04-20 (Actual)

PRIMARY OUTCOMES:
Peak cough flow | baseline
  Peak coughing velocity of voluntary cough in liter/second

SECONDARY OUTCOMES:
Respiratory muscle force | baseline
  MIP/MEP in cmH2O
Pulmonary function test | baseline
  PEF/MVV in liter/min
Pulmonary function test | baseline
  FEV1/FVC/VT in liter
Pulmonary function test | baseline
  MVV rate in breaths/min
Muscle thickness during voluntary force | baseline
  tRA/tEO/tIO/tTrA/tD in millimeter
Muscle activation during voluntary force | baseline
  aURA/aLRA/aEO/aIOTrA/aD (all the data will be collected through surface EMG and will be presented as maximal voluntary contraction in %)
Diaphragm assessment | baseline
  QB_ex/DB_ex/Sniff_ex in millimeter
Diaphragm assessment | baseline
  QB_slope/DB_slope/Sniff_slope in cm/s

CONTACTS AND LOCATIONS:
Overall Officials: Ching-Hsia Hung, PhD, Principal Investigator — Department of physical therapy, National Cheng Kung University
Locations (1):
- National Cheng Kung University Hospital, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mesquita Montes A, Maia J, Crasto C, de Melo CA, Carvalho P, Santos R, Pereira S, Vilas-Boas JP. Abdominal muscle activity during breathing in different postures in COPD "Stage 0" and healthy subjects. Respir Physiol Neurobiol. 2017 Apr;238:14-22. doi: 10.1016/j.resp.2017.01.001. Epub 2017 Jan 7. PMID 28082171
- [Background] Mesquita Montes A, Crasto C, de Melo CA, Santos R, Pereira S, Vilas-Boas JP. The effect of inspiratory and expiratory loads on abdominal muscle activity during breathing in subjects "at risk" for the development of chronic obstructive pulmonary disease and healthy. J Electromyogr Kinesiol. 2017 Jun;34:50-57. doi: 10.1016/j.jelekin.2017.03.005. Epub 2017 Mar 31. PMID 28399443